CLINICAL TRIAL: NCT05152511
Title: Management of Post-circumcision Ischemia
Brief Title: Management of Post-circumcision Ischemia Using Hyperbaric Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Magdy, Principal Investigator, Aswan University Hospital
Other Study IDs: AswanUH3
Record Dates: First submitted 2021-11-14; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Post-circumsion Complications
Keywords: Glans necrosis,; Hyperbaric oxygen,; Male Circumcision,; Pentoxifylline,; Monopolar cautery.
MeSH Terms: interventions — Hyperbaric Oxygenation; Pentoxifylline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All male children who had penile ischaemia after circumcision were included in the study: It is a cohort prospective study. All male children who had penile ischaemia after circumcision were included in the study between April 2017 and October 2020.
  Interventions: Combination Product: Hyperbaric oxygen therapy

INTERVENTIONS:
Combination Product: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy is a specially designed cabinet for infants and neonates with a barometric pressure equal to 760 mmHg for 20 minutes daily, then gradually increase up to one hour daily for 5 days per week (fig. 1). The chamber was kept warm. The babies were fed before entering the chamber and if signs of hunger appear during therapy. The baby was continuously monitored with pulse oximeter. Older children are managed in the conventional Hyperbaric oxygen chamber with the same regimen.
  Other Names: Pentoxifylline

SUMMARY:
Background: Post-circumcision penile ischaemia is a rare but destructive complication. Our goal is to present our experience in the management of children, who had different forms of penile ischaemia, complicating the routine ritual male circumcision.

Material and Methods: All male children who had post-circumcision penile ischaemia between April 2017 and October 2020 were included in the study. A special designed protocol for management of all cases includes a combination of early Pentoxifylline intervenes infusion with Hyperbaric Oxygen inhalation, early catheterization, and appropriate surgical debridement. Data were analyzed inclusively to patient age, the anesthesia method used, Monopolar diathermy usage, early presentation, method of circumcision and positive wound culture.

DETAILED DESCRIPTION:
It is a cohort prospective study. All male children who had penile ischaemia after circumcision were included in the study between April 2017 and October 2020. A special designed protocol includes early admission of a child in Paediatric intensive care unit (PICU). Catheterization by suitable size silicon Foley's catheter appropriate for the age. IV Pentoxifylline in a dose of 10 mg/kg/day divided into 3 equal doses with good monitoring of its side effects mainly tachycardia and convulsions. IV 3rd generation cephalosporin with suitable doses according to the age and body weight. Hyperbaric Oxygen therapy is a specially designed cabinet for infants and neonates with a barometric pressure equal to 760 mmHg for 20 minutes daily, then gradually increase up to one hour daily for 5 days per week (fig. 1). The chamber was kept warm. The babies were fed before entering the chamber and if signs of hunger appear during therapy. The baby was continuously monitored with pulse oximeter. Older children are managed in the conventional Hyperbaric Oxygen chamber with the same regimen. Proper surgical debridement together with daily topic dressing with nitroglycerin ointment (2%). The treatment continued through the admission period. Follow up period range from 6 months up to 3 years.

Data were analyzed inclusively to patient age, the type of medical provider who performed the circumcision, the technique of male circumcision, the anesthesia method used, if any Monopolar diathermy usage, wound suturing after MC, the duration of between male circumcision and presentation to our protocol, and the final condition of the patient at discharge and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

- male children complained of penile ischaemia after circumcision.

Exclusion Criteria:

* other post-circumcision complication not include penile ischaemia
* patients with chronic diseases.

Ages: 1 Month to 6 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — All male children who had penile ischaemia after circumcision were included in the study between April 2017 and October 2020.
Study Population: Twenty-three male children with penile ischaemia from 3076 post-circumcisions complicated patients.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
post-circumcision complication | April 2017 and October 2020
  early and late complication

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Abdelmohsen, Principal Investigator — Aswan University
Locations (1):
- Sarah Magdy Abdelmohsen, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided